CLINICAL TRIAL: NCT02904135
Title: Collection of Circulating Tumor Cells From the Peripheral Blood of Metastatic Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: MiCareo Taiwan Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MBC 2.7
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Circulating Tumor Cells (CTCs)
Keywords: Circulating Tumor Cells
MeSH Terms: conditions — Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- first stage: During the first stage, the patient's baseline blood sample will be mainly used for validating and troubleshooting our instrument with clinical samples.
- second stage: During the second stage, 40 patients will be followed for up to three years after their baseline blood draw to obtain data on their survival status. The CTC results and follow-up data obtained from these samples will help to analyze any correlation with the patient's clinical outcome and further validate the prognosis ability of MiCareo's CTC platform for mBC patients.

SUMMARY:
To address the challenges of isolating and analyzing rare cells, this study aims to validate the instrumentation, the test protocols, and the analysis of patient's outcome to show the instrument's capability to reproducibly and accurately detect CTCs in cancer patients. In order to facilitate the validation process, investigators will only focus on metastatic patients for whom CTCs supposedly present at higher abundance. Investigators propose to enroll cohorts of metastatic breast cancer patients. Blood samples will be collected from these patients before they start any new line of therapy as determined by their doctors. The specific aims are to isolate, enumerate and analyze the number and/or molecular information of circulating tumor cells in patient blood using microfluidic chip-based sorting, imaging, and molecular profiling techniques. Investigators will use this study to optimize diagnostic instrumentation, test blood processing protocols and CTC analysis algorithm. During this study investigators will collect patients' clinical information related to cancer, as well as the patients' survival status to validate the system's prognosis ability.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed written informed consent before enrollment into the study, ability to communicate with the investigators, and to understand and comply with the requirements of the study.
2. Progressive and measurable metastatic breast cancer.
3. Commencement of new anti-cancer chemotherapy or palliative care.
4. ECOG performance status equal or less than grade 2.

Exclusion Criteria:

1. Subject has received any investigational agent, not explicitly approved by MiCareo, within last one year.
2. Subject being identified with any blood borne infectious disease.
3. Subject has received anticancer chemotherapy within last one month. (not including hormone therapy, or target therapy)
4. Pregnancy.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: metastatic breast cancer (mBC) patients
Sampling Method: Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2014-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Overall survival(OS) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Chen Jui-Lin, Study Director — CEO
Locations (1):
- Keelung Chang Gung Memorial Hospital, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided